CLINICAL TRIAL: NCT04528797
Title: Cadaveric Organ Donor Management: Thyroid and Adrenocortical Hormone Replacement
Brief Title: Thyroid and Adrenocortical Hormone Replacement in Organ Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: We Are Sharing Hope SC (Unknown)
Responsible Party: Principal Investigator, Adrian Van Bakel, Professor of Medicine, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR 17718
Record Dates: First submitted 2020-08-20; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Brain Death
MeSH Terms: conditions — Brain Death | interventions — Thyroxine; Methylprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Levothyroxine (Experimental): Levothyroxine 20 mcg IV bolus initiated at the beginning of active donor management followed by continuous infusion of 50 to 200 mcg/hr titrated to minimize vasopressor requirements until organ procurement.
  Interventions: Drug: Levothyroxine
- Methylprednisolone (Experimental): Methylprednsiolone 30 mg/kg (up to 2 g) IV initiated at the beginning of active donor management followed by repeat dosing of 15 mg/kg (up to 1 g) 12 hours later.
  Interventions: Drug: Methylprednisolone
- Combination (Experimental): Methylprednsiolone 30 mg/kg (up to 2 g) IV initiated at the beginning of active donor management followed by repeat dosing of 15 mg/kg (up to 1 g) 12 hours later plus levothyroxine 20 mcg IV bolus initiated at the beginning of active donor management followed by continuous infusion of 50 to 200 mcg/hr titrated to minimize vasopressor requirements until organ procurement.
  Interventions: Drug: Levothyroxine; Drug: Methylprednisolone
- Control (No Intervention): No levothyroxine or methylprednisolone administered.

INTERVENTIONS:
Drug: Levothyroxine
  Arms: Combination; Levothyroxine
Drug: Methylprednisolone
  Arms: Combination; Methylprednisolone

SUMMARY:
Brain death inevitably leads to hemodynamic instability and prolonged hypotension that compromises viability of potentially transplantable organs. In addition to depletion of peripheral norepinephrine stores, concomitant depletion of thyroid hormone and cortisol levels are believed to contribute to this instability. Catecholamine vasopressors are widely used to support hemodynamics in potential organ donors, however their use has also been shown to compromise allograft function.

Trials studying the effects of thyroid hormone and corticosteroid treatment on brain dead organ donors have had mixed results with respect to improving donor hemodynamics. Further, few studies have attempted to discriminate the relative contribution of thyroid hormone vs. corticosteroids.

The specific aims of this study include:

1. To quantify hemodynamic changes during the management of cadaveric organ donors routinely receiving thyroid hormone therapy alone vs. corticosteroid therapy alone vs. the combination, compared to those who do not receive any hormonal therapy (controls)
2. To document number and types of organs procured in donors treated with thyroid hormone therapy alone vs. corticosteroid therapy alone vs. the combination, compared to those not treated with hormonal therapy (controls)
3. To quantify graft and patient outcomes in recipients of organs exposed to thyroid hormone therapy alone vs. corticosteroid therapy alone vs. the combination, compared to recipients of organs not exposed to hormonal therapy (controls).

ELIGIBILITY:
Inclusion Criteria:

Cadaveric organ donors ≥ age 18 having valid consent (by advance directive or by familial consent) to donate organs.

Recipients of these cadaveric organs

Exclusion Criteria:

Cadavers failing to meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2010-09-02 (Actual); Primary Completion 2012-08-09 (Actual); Study Completion 2013-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Vasoactive Inotrope Score (VIS) score from beginning of active donor management until procurement. | From baseline (t0) = beginning of active donor management to procurement (tOR) = time of organ procurement, up to 50 hours
  The VIS score includes all commonly used vasopressor and inotrope agents, weighted by potency and summed

SECONDARY OUTCOMES:
Proportion of organs procured vs. consented, stratified by treatment group | assessed at time of procurement, up to 50 hours following consent for donation
Recipient Morbidity | 90 days post transplant
  Selected graft recipient morbidity measures in all organs transplanted stratified by treatment group
Recipient Mortality | 90 days post traansplant
  Recipient death by 90 days post transplant

IPD SHARING:
Plan to Share IPD: No
There is currently no plan in place to share IPD for this study

REFERENCES:
- [Derived] Van Bakel AB, Hino SA, Welker D, Morella K, Gregoski MJ, Craig ML, Crumbley AJ, Sade RM. Hemodynamic Effects of High-dose Levothyroxine and Methylprednisolone in Brain-dead Potential Organ Donors. Transplantation. 2022 Aug 1;106(8):1677-1689. doi: 10.1097/TP.0000000000004072. Epub 2022 Jul 22. PMID 35389961